CLINICAL TRIAL: NCT02812862
Title: Cardiac Effects of Spiolto®/Respimat® in Patients With Congestive Heart Failure and COPD
Acronym: CREATES
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Rationale obsolete
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-165
Record Dates: First submitted 2016-06-14; First posted 2016-06-24 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): 20 male and female patients suffering from chronic heart failure and chronic obstructive pulmonary disease.
  Patients will be treated with Spiolto® Respimat® (the LABA/ LAMA combination)
  Interventions: Drug: Spiolto® Respimat® (Tiotropium / Olodaterol)

INTERVENTIONS:
Drug: Spiolto® Respimat® (Tiotropium / Olodaterol) — LABA/ LAMA combination therapy:
  A combination of two bronchodilators acting on two separate pharmacological targets - one ß-agonist and one anti-muscarinergic agent.
  Other Names: Long-acting ß-agonist (LABA); Long-acting anti-muscarinergic agent (LAMA)

SUMMARY:
The aim of this study is to evaluate the pulmonary and cardiac effects of the LABA / LAMA combination Tiotropium / Olodaterol therapy in patients suffering from both congestive heart failure and chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are contractually capable and mentally able to understand and follow the instructions of the study personnel
* Symptomatic with regard to dyspnea (NYHA II-III, mMRC Dyspnea score > 1)
* Diagnosis of COPD (FEV1/FVC ratio <70%, FEV1 < 80%)
* Patients with hyperinflation at rest defined as Residual Volume (RV) > 135 % predicted
* Diagnosis of moderate symptomatic ischaemic Congestive heart failure (LVEF > 35 -45%)
* Stability of CHF during the preceding 3 months (no hospitalization due to CHF, stable CHF medication)
* Male or female aged > 18 years
* Written informed consent prior to study participation
* The subject is willing and able to follow the procedures outlined in the protocol

Exclusion Criteria:

* Lack of informed consent
* Pregnant and lactating females
* Acute moderate-severe exacerbation of COPD, acute respiratory failure (pH < 7,35 and/ or respiratory rate > 30/min within 3 months prior to inclusion)
* Unstable heart failure or planned change in medication (hospitalization due to CHF within 3 months prior to inclusion), any angina pectoris
* Not symptomatic
* Patient has been committed to an institution by legal or regulatory order
* Participation in a parallel interventional clinical trial
* Any COPD maintenance therapy before start of randomization
* History or diagnosis of Asthma
* LVEF <35 % or ICD or pacemaker
* Myocardial infarction 6 months prior inclusion
* History of life-threatening arrhythmias (e.g. NSVT or ventricular tachycardia, aFib, AV-Block, pacemaker treatment etc.)
* History of diagnosis of Thyrotoxicosis
* Chronic kidney disease with an crea-clearance ≤30 ml/min
* History of significant alcohol or drug abuse, as judged by the Investigator
* Fibrotic lung disease (e.g. IPF, ILD)
* Contraindications for MRT (e.g. pacemaker, defibrillator, ferromagnetic metal implants, tattoos, claustrophobia, etc. according to MRI checklist used in the clinical routine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
To examine the change in Residual Volume (RV) V0-V2 | 24 months

SECONDARY OUTCOMES:
To examine the change in trough FEV1 | 24 months
  Time Points: values at V0 compared with V2

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, MD, Principal Investigator — University Hospital, Aachen
Locations (1):
- Clinic of Cardiology, Angiology, Pneumology and Intensive Medicine, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bateman ED, Ferguson GT, Barnes N, Gallagher N, Green Y, Henley M, Banerji D. Dual bronchodilation with QVA149 versus single bronchodilator therapy: the SHINE study. Eur Respir J. 2013 Dec;42(6):1484-94. doi: 10.1183/09031936.00200212. Epub 2013 May 30. PMID 23722616
- [Background] Dahl R, Chapman KR, Rudolf M, Mehta R, Kho P, Alagappan VK, Chen H, Banerji D. Safety and efficacy of dual bronchodilation with QVA149 in COPD patients: the ENLIGHTEN study. Respir Med. 2013 Oct;107(10):1558-67. doi: 10.1016/j.rmed.2013.05.016. Epub 2013 Jul 16. PMID 23867808